CLINICAL TRIAL: NCT04229420
Title: Comparison of Ultrasound-Guided Bilateral Erector Spinae Plane Block Versus Bilateral Rectus Sheath Block in Adults Undergoing Major Abdominal Surgery: a Randomized Comparative Study.
Brief Title: Comparison of Ultrasound-Guided Bilateral Erector Spinae Plane Block Versus Bilateral Rectus Sheath Block in Adults Undergoing Major Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, principal investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MD-33-2019
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Pain; Postoperative
Keywords: erector spinae; ultrasound; rectus sheath; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Study will be conducted on 60 adults aged from 18 to 60 years presented for major abdominal surgeries (open colorectal resections or major ventral hernia repair) at general surgery operating theatres, Cairo university hospitals.
  Patients will be divided into two equal groups; rectus sheath block group RSB (n=30) and erector spinae plane block group ESPB (n=30).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectus sheath block group (RSB) (Active Comparator): After preparing the skin, a high frequency (5-10 MHz) ultrasound probe will be placed in a longitudinal orientation above the level of the umbilicus with the Patient in the supine position. After identifying the rectus abdominis muscle, A 22 G echogenic needle using the in plane technique will be inserted just below the costal margin then, a total of 20 ml of 0.25% bupivacaine will be injected into the plane between the rectus muscle and posterior rectus sheath. Negative aspiration will be confirmed every 5 ml. The block will then be repeated on the other side.
  Interventions: Device: Ultrasound guided Rectus sheath block vs Erector spinae plane block
- Erector spinae plane block group (ESPB) (Active Comparator): After induction of anesthesia; the patient will be positioned on the lateral position. The skin will be prepared with povidone iodine, and a high frequency (5-10 MHz) ultrasound probewill be placed in a transverse orientation on the T9 spinous process which will be located by palpating and counting down from the C7 spinous process. The tip of the T9 transverse process will be identified and centred on the ultrasound screen, the probe will then be rotated into a longitudinal orientation to produce a parasagittal view. Correct location of the needle tip in the fascial plane deep to erector spinae muscle is conﬁrmed by injecting 0.5-1 ml saline and seeing the ﬂuid lifting the erector spinae muscle off the transverse process while not distending the muscle. A total of 20 ml of 0.25% bupivacaine will then be injected into the ESP of both sides.
  Interventions: Device: Ultrasound guided Rectus sheath block vs Erector spinae plane block

INTERVENTIONS:
Device: Ultrasound guided Rectus sheath block vs Erector spinae plane block — Ultrasound guided Rectus sheath block vs Erector spinae plane block

SUMMARY:
This randomized, controlled study is designed to assess the quality of analgesia provided by ultrasound guided ESPB versus RSB in adults undergoing major abdominal surgery.

DETAILED DESCRIPTION:
Introduction:

Regional anesthesia is a key component of opioid-sparing multimodal analgesia after major abdominal surgery as it improves recovery such as return of bowel function and early ambulation. Continuous epidural local anesthetic infusion is a common analgesic technique but comes with the side effect of hypotension and potential leg weakness and rarely, epidural abscess or hematoma. The rectus sheath block (RSB) has been used for postoperative analgesia in surgical procedures involving a vertical midline laparotomy incision as well as for laparoscopic procedures. In this block the ventral rami of the seventh intercostal nerve up to the subcostal nerve, which supply the rectus abdominis muscle and overlying skin, are blocked.

Recently, the erector spinae plane block (ESPB) has gained wide attention due to its simplicity and potential uses in truncal procedures. This paraspinal plane block is performed by injecting local anesthetic between the erector spinae muscles and transverse processes and is thought to work by blocking the dorsal and ventral rami of the thoracic spinal nerves. Injections at various thoracic levels have been described in case reports with satisfactory postoperative analgesia for breast, thoracic and abdominal procedures. Comparison of post-operative pain management of both erector spinae plane block and rectus sheath block in adults undergoing major abdominal surgery for has not been investigated before.

Hypothesis:

It is hypothesized that ESPB is more effective in postoperative analgesia following major abdominal surgeries with minimal motor affection and postoperative morphine consumption compared to RSB block.

2. Study Protocol:

On arrival of the patients to anesthesia room, patients will be secured with 20-gauge intravenous cannula and will receive midazolam 0.02mg/kg intravenous (IV), ondansetron (4 mg slowly IV).

Monitoring will include ECG, non-invasive arterial blood pressure, and pulse oximetry (SpO2).

All patients will receive a standardized anesthetic technique for induction with 2mcg/kg fentanyl, 2-3 mg/kg propofol, and 0.5 mg/kg atracurium. Mechanical ventilation will be adjusted to maintain an end tidal CO2 between (30 - 40 mmHg). Maintenance will be achieved with oxygen/air with isoflurane 1.2% and atracurium infusion at a dose of 0.5 mg/kg/h.

Following induction of anesthesia patients will be divided into two equal groups; Group 1 will receive pre-incisional ultrasound (US)-guided Bilateral RSB blocks using 20-ml volume of bupivacaine 0.25% for each side, and group 2 will receive pre-incisional ultrasound (US)-guided Bilateral ESPB using 20-ml volume of bupivacaine 0.25% for each side.

Group 1(RSB):

After preparing the skin with povidone iodine, a high frequency (5-10 MHz) ultrasound probe (S-NerveTM; SonoSite Inc., Bothell, WA, USA) will be placed in a longitudinal orientation above the level of the umbilicus with the Patient in the supine position. After identifying the rectus abdominis muscle, A 22 G echogenic needle using the in plane technique will be inserted just below the costal margin at an angle of approximately 45 degrees to the skin, then, a total of 20 ml of 0.25% bupivacaine will be injected into the plane between the rectus muscle and posterior rectus sheath. Negative aspiration will be confirmed every 5 ml. The block will then be repeated on the other side.

Group 2 (ESPB):

After induction of anesthesia; the patient will be positioned on the lateral position. The skin will be prepared with povidone iodine, and a high frequency (5-10 MHz) ultrasound probe (S-NerveTM; SonoSite Inc., Bothell, WA, USA) will be placed in a transverse orientation on the T9 spinous process which will be located by palpating and counting down from the C7 spinous process. The tip of the T9 transverse process will be identified and centred on the ultrasound screen, the probe will then be rotated into a longitudinal orientation to produce a parasagittal view, visible superﬁcial to the acoustic shadows of the transverse processes: skin and subcutaneous tissue; trapezius; and erector spinae muscle .Correct location of the needle tip in the fascial plane deep to erector spinae muscle is conﬁrmed by injecting 0.5-1 ml saline and seeing the ﬂuid lifting the erector spinae muscle off the transverse process while not distending the muscle. A total of 20 ml of 0.25% bupivacaine will then be injected into the ESP of both sides. Negative aspiration will be confirmed every 5 ml].

Postoperative pain management:

Postoperatively, patients will receive 1 g paracetamol every 6 h and 30 mg ketorolac every 12 h.

If the visual analogue scale (VAS) is ≥ 4, a morphine increment (2-3 mg) IV that could be repeated every 5 minutes with a maximum dose of 15 mg per 4 hours or 45 mg per 24 hours will be added to maintain a resting VAS at <4 and the total 24 hours morphine consumption will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II. Age: 18 to 60 years. Undergoing midline vertical laparotomy incisions (open colorectal resections or major ventral hernia repair).

Exclusion Criteria:

1. Refusal of patients.
2. Patients with coagulation disorders (Platelets ≤ 50,000 and/or INR> 1.5).
3. History of allergic reactions to local anesthetics.
4. Rash or signs of infection at the injection site.
5. Emergency surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Time to first request of postoperative rescue analgesics | 24 hours
  the time interval between the block performance and the first request to postoperative analgesia and or VAS ≥ 4

SECONDARY OUTCOMES:
Visual analogue score at rest (static), and on movement or coughing (dynamic) | 24 hours
  Visual analogue score at rest (static), and on movement or coughing (dynamic) at 30 and 60 minutes in the PACU then every 6 hours in the ward for 24 hours.
  The visual analogue score is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length.
  For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale])
Total consumption of morphine | 24 hours
  total postoperative morphine consumption
Incidence of perioperative complications. | 24 hours
  Incidence of perioperative complications(lower limb weakness, hematoma, viscus injury, intravascular injection and PONV
Block performance time in min | procedure (time from probe contact with skin till needle withdrawal)
  time from probe contact with skin till needle withdrawal.
Failure rate of the block | 1st postoperative hour
  will be calculated, where the block will be considered a failed block if the patient required more than two doses of rescue analgesia in the first hour postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Sarhan, MD, Principal Investigator — Lecturer of anesthesia, Cairo university
Locations (1):
- Kasralainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided